CLINICAL TRIAL: NCT04624386
Title: Evaluating Oxidative Stress in Postmenopausal Women
Brief Title: Evaluating Oxidative Stress in Menopause
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nura Fitnat Topbas Selcuki, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: menopausethiol
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Menopause; Oxidative Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thiol disulfide level in venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal/Study: Women older than 45 years of age and who have not had any menstruation for the past 12 months are considered as having entered menopause. These women are included in this group.
  Interventions: Other: Thiol disulfide level
- Premenopausal/Control: Healthy women who are still having regular menstruations are included in this group
  Interventions: Other: Thiol disulfide level

INTERVENTIONS:
Other: Thiol disulfide level — Venous blood is collected from all subjects and thiol disulfide levels will be determined from the serum samples obtained from the venous blood.

SUMMARY:
Thiol disulfide levels will be determined using venous blood samples from pre- and postmenopausal women to evaluate oxidative stress in menopause. Furthermore, oxidative stress will be assessed according to age, and years since the start of menopause. Also, whether the presence of menopause related osteoporosis has any association with oxidative stress will be determined.

DETAILED DESCRIPTION:
A total of 77 subjects are divided into two groups: study group (postmenopausal women) and control group premenopausal women). Biometric data such as age, bmi, obstetric anamnesis, history of komorbidities, PAP smear results are recorded. Mammography results, dexa scores of post menopausal women are also obtained. Venous blood samples from all subjects are collected. Thiol disulfide levels will be determined from serum samples. Thiol disulfide levels will first be compared between the study and the control group in order to determine the oxidative stress in menopause. In secondary evaluation years of menopause, age, and dexa scores will be included.

ELIGIBILITY:
Inclusion Criteria:

Women who entered menopause as a natural process Women within the age limits Still menstruating healthy women as control subjects

Exclusion Criteria:

Women who have entered menopause prematurely Women who have entered menopause following a surgery Women with medically induced menopause Women without any autoimmune or chronic inflammatory diseases Women who are taking hormone replacement therapy due to menopausal symptoms Women without any malignant diseases

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women within 30-75 years of age were recruited to this study. Premenapusal healthy women who visited the clinic for routine gynecological control were included in the control group. Postmenopausal women older than 45 years of age who entered menopause as a natural process were included in the study group.
  A total of 43 subjects were included in the study group and 34 subjects were included in the control group
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Evaluating Oxidative Stress in Menopause | 2 months
  Thiol disulfide stress will be evaluated using serum samples from postmenopausal women and comparing these results with samples obtained from premenopausal women.

SECONDARY OUTCOMES:
Evaluating Oxidative Stress According to Years of Menopause | 2 months
  Thiol disulfide levels will be determined and analysis will be done according to the years of menopause
Evaluating Oxidative Stress According to Menopause Related Osteoporosis | 2 months
  Thiol disulfide levels will be determined and analysis will be done according to the osteoporosis scores evaluated with dxa

CONTACTS AND LOCATIONS:
Overall Officials: Nura Fitnat Topbas Selucki, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No